CLINICAL TRIAL: NCT06527287
Title: Neurocognitive Ankle Training for Instability to Optimize Neuromusculoskeletal Outcomes (NATION)
Acronym: NATION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Megan Roach, Musculoskeletal Health Researcher, Womack Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-19385; MO240042 (Other Grant/Funding Number: MOMRP)
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Ankle Instability
Keywords: Chronic Ankle Instability; neurocognition; evidence-based rehabilitation; musculoskeletal outcomes; dual tasks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NATION (Experimental): NATION is a 6-week evidence-based CAI rehabilitation protocol that incorporates neurocognitive exercises. Participants will complete 18 unsupervised home sessions and 12 supervised sessions over the course of 6-weeks.
  Interventions: Other: Neurocognitive Ankle Training for Instablity to Optimize Neuromusculoskeletal outcomes (NATION)
- Evidence-based (Active Comparator): The Evidence-Based protocol will be identical to the intervention (i.e., NATION protocol), but the exercises will exclude the neurocognitive tasks. Participants will complete 18 unsupervised home sessions and 12 supervised sessions over the course of 6-weeks.
  Interventions: Other: Evidence-Based
- Control (No Intervention): Participants assigned to the Control arm will be instructed to continue their normal routine.

INTERVENTIONS:
Other: Neurocognitive Ankle Training for Instablity to Optimize Neuromusculoskeletal outcomes (NATION) — The NATION rehabilitation protocol will serve as the true intervention group. NATION is a 6-week evidence-based chronic ankle instability (CAI) rehabilitation protocol that incorporates neurocognitive exercises. Participants will complete up to 18 unsupervised home sessions and up to 12 supervised sessions. Treatment volume and exercises may vary based on participant progress and study team member guidance.
  Arms: NATION
Other: Evidence-Based — The Evidence-Based rehabilitation protocol will serve as the active comparator group. The Evidence-Based protocol will be similar to the intervention (i.e., NATION protocol), but the exercises will exclude the neurocognitive tasks. Participants assigned to the Evidence-Based protocol will complete up to 18 unsupervised home sessions and up to 12 supervised sessions over the course of 6-weeks. Treatment volume and exercises may vary based on participant progress.
  Arms: Evidence-based

SUMMARY:
The purpose of this study is to examine the effectiveness of a novel ankle rehabilitation protocol on improving clinical and health outcomes in physically active individuals with chronic ankle instability (CAI). Our central hypothesis is NATION, a novel rehabilitation intervention that includes neurocognitive tasks, will improve overall health and function, and reduce lower extremity musculoskeletal injury in physically active individuals with CAI.

DETAILED DESCRIPTION:
Military personnel and physically active civilians are particularly vulnerable to ankle sprains and subsequent chronic ankle instability (CAI). CAI is a complex neuromusculoskeletal condition characterized by recurring ankle sprains, episodes of instability, ongoing pain, and functional disability that results in activity limitations and participation or duty restrictions. Despite mitigation efforts, ankle sprains continue to occur frequently and commonly progress to CAI.

CAI is associated with deficiencies in neurocognitive function (i.e., the ability to think, reason, and react) and increased instability during dual-tasks. These neurocognitive deficiencies identify a novel impairment that should be addressed during CAI rehabilitation. However, current evidence-based protocols for CAI lack dual-task exercises that incorporate visual and cognitive components simultaneously. Thus, training neurocognitive function simultaneously with traditional CAI impairments, may improve outcomes and mitigate episodes of giving way, recurrent ankle sprains, and subsequent lower extremity Musculoskeletal Injuries (MSKIs), culminating in improved Service member and civilian outcomes, continued involvement in physical activity, and active duty status retention. Hence, the overall objective of the Neurocognitive Ankle Training for Instability to Optimize Neuromusculoskeletal outcomes (NATION) study, is to examine the effectiveness of a novel ankle rehabilitation protocol on improving clinical and health outcomes in physically active individuals with CAI.

The overall objective will be achieved by the following Specific Aims:

Specific Aim 1: Determine the effectiveness of NATION on improving clinical outcomes compared to an evidence-based rehabilitation intervention and control arm in physically active individuals with CAI at 6-weeks and 6-months post-enrollment.

Hypothesis 1: Our novel CAI rehabilitation protocol will result in improved range of motion, postural control, strength, somatosensation, lower extremity function, and motor-cognition as compared to an evidence-based protocol and control arm.

Specific Aim 2: Determine the effectiveness of NATION on improving health outcomes compared to an evidence-based rehabilitation intervention and control arm in physically active individuals with CAI at 6-weeks and 6-months post-enrollment.

Hypothesis 2: Our novel CAI rehabilitation protocol will result in improved self-reported function and quality of life, less injury-related fear and pain, fewer episodes of the ankle giving way, and lower MSKI rates compared to an evidence-based protocol and control arm.

Specific Aim 3: Determine the effectiveness of NATION on improving Service member outcomes compared to an evidence-based rehabilitation intervention and control arm in Service members with CAI at 6-weeks and 6-months post-enrollment.

Hypothesis 3: Our novel CAI rehabilitation protocol will result in improved confidence to deploy compared to an evidence-based protocol and control arm.

Specific Aim 4: Determine the effectiveness of NATION on reducing surgical intervention rates compared to an evidence-based rehabilitation intervention and control arm in Service members with CAI up to 60-months post-enrollment.

Hypothesis 4: Our novel CAI rehabilitation protocol will result in fewer Service members requiring surgical intervention for CAI within 60-months compared to an evidence-based protocol or control arm.

Specific Aim 5: Compare participant workload (mental, physical, temporal, performance, effort, frustration) over time and between intervention arms.

Hypothesis 5: The participants' perception of workload will gradually increase from Week 1 to Week 6 and NATION participants will perceive an increased workload compared to the evidence-based participants.

Specific Aim 6: Assess participant satisfaction with the NATION and evidence-based rehabilitation programs.

Hypothesis 6: Our novel CAI rehabilitation protocol will result in improved satisfaction compared to an evidence-based protocol intervention.

This is a multi-site single-blind randomized controlled trial to determine the effectiveness of NATION on improving clinical (Specific Aim #1), health (Specific Aim #2), and Service member (Specific Aim #3) outcomes, and reducing the need for surgical intervention (Specific Aim #4) in individuals with CAI. Participant workload throughout the NATION and Evidence-Based Practice interventions (Specific Aim #5) and participant satisfaction with the rehabilitation interventions (Specific Aim #6) will also be assessed.

The study includes two unique rehabilitation protocols (NATION and Evidence-Based) and a Control group. Participants will be randomized to one of the three treatment groups: (1) NATION, (2) Evidence-Based Rehabilitation, or (3) No Treatment. A study team member blinded to treatment group will collect the outcome measures. An unblinded study team member will reveal the participant's treatment group and conduct the NATION and Evidence-Based rehabilitation sessions.

The NATION rehabilitation protocol will serve as the true intervention group. NATION is a 6-week evidence-based CAI rehabilitation protocol that incorporates neurocognitive exercises. Participants will complete up to 18 unsupervised home sessions and up to 12 supervised sessions. Supervised sessions will be conducted up to 2 times per week and will include evidence-based range of motion, strength, and balance exercises as well as plantar massage for the involved ankle. The Evidence-Based rehabilitation protocol will serve as the active comparator group. The protocol will be identical to the intervention (i.e., NATION protocol), but the exercises will exclude the neurocognitive tasks. Participants assigned to the Evidence-Based protocol will complete up to 18 unsupervised home sessions and up to 12 supervised sessions over the course of 6-weeks. Participants assigned to no treatment will be instructed to continue their normal routine.

Study participants will complete clinical and health outcome assessments upon enrollment and 6-weeks and 6-months post-enrollment. Only active-duty Service members will complete the Service member outcome assessments upon enrollment, 6-weeks and 6-months post-enrollment. For Specific Aim #1, all participants will complete: 1) dorsiflexion range of motion via the Weight Bearing Lunge Test; 2) ankle strength assessments in all four planes utilizing a hand-held dynamometer; 3) dynamic and static balance assessments utilizing the Star Excursion Balance Test and force plate measures; 4) somatosensation utilizing the Semmes Weinstein Monofilament 4-2-1 stepping algorithm; and 5) motor-cognitive assessments including a Choice-Reaction Hop-to-Stabilization Task and a Lower Extremity Reaction Time Task. Clinical outcomes will be collected upon enrollment (i.e., baseline), 6-weeks, and 6-months post-enrollment. For Specific Aim #2, all participants will complete: 1) self-reported measures of pain, fear, function, and physical activity including the Cumberland Ankle Instability Tool, Defense and Veterans Pain Rating Scale, Fear-Avoidance Beliefs Questionnaire, Modified Disablement in the Physically Active Scale, the National Aeronautics and Space Administration (NASA) Physical Activity Scale, and the Quick-Foot and Ankle Ability Measure; and 2) self-reported MSKI history/new MSKI during the study follow-up period. Health outcomes will be collected upon enrollment (i.e., baseline), 6-weeks, and 6-months post-enrollment. For Specific Aim #3, all active-duty Service members participating will complete a self-reported measure of confidence to deploy. Confidence to deploy will be collected upon enrollment (i.e., baseline), 6-weeks, and 6-months post-enrollment. For Specific Aim #4, all Defense Enrollment Eligibility Reporting System (DEERS) eligible participants medical records will be actively surveilled for surgical interventions related to CAI for up to 60-months post-enrollment. For Specific Aim #5, all participants assigned to NATION or the Evidence-Based Practice rehabilitation intervention will complete the NASA Task Load Index following each supervised intervention session. For Specific Aim #6, all participants assigned to NATION or the Evidence-Based Practice rehabilitation intervention will complete a self-reported patient satisfaction questionnaire upon completion of treatment.

To address Specific Aims 1, 2, and 3 an analysis of covariance (ANCOVA)-type linear mixed effect (LME) model will be used to model the data. The fixed effects of the LME model will be intervention (NATION, Evidence-Based, Control), sex, and time, along with all 3-way (group*sex*time), as well as 2-way (group*sex, group*time, sex*time) interaction effects of these variables. The random effects of the LME model will be participant-specific intercepts and slopes. To account for missingness due to dropout or lack of follow-up we will employ an intention-to-treat analysis strategy.

For Specific Aim 4, the response variable will be time-to-surgical intervention along with the binary event status indicator (non-responder=1, responder=0). For participants who go on to have ankle surgery (non-responders), the time elapsed in days between enrollment and the surgery date will be recorded for the event time. For participants who do not go on to have ankle surgery (responder), the censoring time will time from enrollment to the end of the surveillance period or time of drop-out/disenrollment (whichever occurs first). To analyze the data, a Cox-regression model will be fit to the data which uses treatment group, sex, and treatment group*sex interaction.

To address Specific Aim #5, participant workload will be compared over time and between intervention arms (NATION vs Evidence-Based) using a two-way repeated measures ANOVA. Both individual workload domains and total scores will be assessed as applicable.

To address Specific Aim #6, participant satisfaction will be compared between intervention arms (NATION vs Evidence-Based). Satisfaction with the overall intervention, duration of treatment, ability to address health issues, and likelihood to recommend the intervention as well as a Total Satisfaction score will be analyzed using Mann-Whitney U-tests or other statistical approach as appropriate for the data.

ELIGIBILITY:
Inclusion Criteria:

* Physically active and engage in regular exercise/training
* 18-44 years old (accounts for 86% of the individuals deployed in recent military conflicts)
* Answer "yes" to Question 1 (i.e., have you ever sprained an ankle?) on the Ankle Instability Instrument
* Answer "yes" to any four of the remaining Ankle Instability Instrument questions
* Score <24 on the Cumberland Ankle Instability Tool
* Report at least two episodes of the ankle "giving way" in the last six months
* Access to a functional email address and internet for completion of health and Service member outcomes
* Ability to provide informed consent

Exclusion Criteria:

* Unable to read or comprehend the English language.
* An ankle sprain within the last six (≤6) weeks that resulted in altered or missed physical activity for one or more (≥1) consecutive days.
* History of ankle surgery.
* History of lower extremity fracture in the last year or history of fracture that required fixation.
* Any peripheral neuropathies or other health conditions/current musculoskeletal injuries that may influence balance.
* Pregnant females (will be eligible for participation in the study after delivery of the baby and medical clearance by a qualified and licensed healthcare provider).

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-14 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Ankle Strength | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Ankle plantarflexion, dorsiflexion, inversion, and eversion peak isometric force will be assessed with a hand-held dynamometer
Balance | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Static and dynamic balance will be captured via a force plate and the Star Excursion Balance Test.
Motor Cognition | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Motor-cognition will be measured via a choice reaction hop-to-stabilization test and a lower extremity reaction time task.
Ankle Range of Motion | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Dorsiflexion range of motion will be measured via the Weight-Bearing Lunge test.
Somatosensation | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Somatosensation will be measured at the center of the heel using the 4-2-1 Semmes-Weinstein monofilament stepping algorithm.

SECONDARY OUTCOMES:
Fear-Avoidance Beliefs Questionnaire | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Injury-related fear will be captured on the ankle-specific Fear-Avoidance Beliefs Questionnaire (FABQ). The FABQ is a 16-item questionnaire designed to assess fear-avoidance beliefs regarding physical activity and work. FABQ total scores range from 0 to 66 with higher scores indicating greater fear.
Quick-Foot and Ankle Ability Measure | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Foot and ankle function will be measured via the Quick Foot and Ankle Ability Measure (Quick-FAAM). A 12-item scale, the Quick-FAAM is comprised of two subscales: Activities of Daily Living (FAAM-ADL) and Sport (FAAM-Sport). All scores are transformed into percentages, with 100% representing no functional loss.
Defense and Veterans Pain Rating Scale | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Quality of life will be assessed via the modified Disablement in the Physically Active Scale (mDPA). The mDPA is a 16-item generic outcome instrument designed by athletic trainers for physically active individuals. The mDPA scores range from 0 to 64 with higher scores indicating greater disablement.
Modified Disablement in the Physically Active Scale | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Quality of life will be assessed via the modified Disablement in the Physically Active Scale (mDPA). The mDPA is a 16-item generic outcome instrument designed by athletic trainers for physically active individuals. The mDPA scores range from 0 to 64 with higher scores indicating greater disablement.
Confidence to Deploy | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Participants will rate their ability to travel to/within a combat zone, carry/wear/use all required equipment and/or weapon, and perform required military duties for the duration of a six month deployment on a scale of 0 (not at all confident) to 100 (fully confident).
Musculoskeletal Injury Questionnaire | Baseline, 6-weeks post-enrollment, & 6-months post-enrollment
  Participants will self-report lifetime ankle sprains and any previous lower extremity MSKIs sustained 12-months prior to enrollment into the study. Participants will also self-report number of episodes of the ankle giving way and any new lower extremity MSKIs at 6-weeks and 6-months post-enrollment.

OTHER OUTCOMES:
NASA Task Load Index | At the completion of each supervised rehabilitation session.
  All six NASA Task Load Index dimensions will serve as an outcome of interest on a scale of 0 (very low) to 100 (very high).
Participant Satisfaction Questionnaire | At the conclusion of the 6-week intervention for participants assigned to the NATION and Evidence-Based Practice protocols.
  To assess participant satisfaction with the interventions participants will complete the Participant Satisfaction Questionnaire. Each question is scored on a Likert scale of 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Megan H Roach, Principal Investigator — Womack Army Medical Center

IPD SHARING:
Plan to Share IPD: No